CLINICAL TRIAL: NCT07185607
Title: Effect of the Erector Spinae Plane Block in Patients Undergoing Robotic Colorectal Surgery
Brief Title: Effect of the Erector Spinae Plane Block in on Robotic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Taner Abdullah, MD, Istanbul Saglik Bilimleri University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-485
Record Dates: First submitted 2025-09-08; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Erector Spinae Plane Block; Robotic Surgery; Postoperative Pain Management; Colorectal Surgery
Keywords: erector spinae plane block; robotic surgery; postoperative pain management; colorectal surgery

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The block was performed with the patients' consent. The control group did not receive the block. Therefore, due to the nature of the procedure, the patients were not blinded.
  The block operator was not blinded.
  The primary investigator assessing the patient outcomes did not know which patients received the block and which did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB + group (Active Comparator): the patients who received ESPB
  Interventions: Procedure: Erector spinae plane block (ESPB)
- ESPB - group (No Intervention): the patients who not received ESPB

INTERVENTIONS:
Procedure: Erector spinae plane block (ESPB) — Erector spinae plane block is not a drug or a device. It is a regional method for anesthesia/analgesia. Before block application, patients were placed in a sitting position. A preliminary examination with a high-frequency linear probe was performed to identify the application site. Sterile conditions were then established. An ultrasound probe was longitudinally placed approximately 2 cm lateral to the T11 spinous process. The transverse process was visualized. 1 ml of 2% lidocaine was applied to the estimated needle entry site. The needle was then guided toward the transverse process using an out-of-plane method using a blocking needle (Stimuplex® Ultra 360® 22G 80 mm, Melsungen, Germany). After bone contact was achieved, facial hydrodissection was observed with 1-2 ml of saline solution to verify the correct injection site. 20 ml of 0.25% bupivacaine was injected into the plane. The distribution of the drug was visualised by USG.
  Arms: ESPB + group

SUMMARY:
The primary objective of this study is to demonstrate whether the Erector Spinae Plane Block provides effective analgesia in patients undergoing robotic colorectal surgery and whether it contributes positively to the postoperative process.

With the advantages of ultrasound in recent years, the application of regional anesthesia methods such as trunk and peripheral nerve blocks has become a crucial component of multimodal analgesia strategies in postoperative pain management. Among regional techniques, the erector spinae plane block, in particular, has been shown to provide effective analgesia after numerous surgeries in recent years and is increasingly being used. Because the erector spinae plane block provides effective analgesia in a wide range of thoracic and abdominal surgeries, such as thoracotomy, cholecystectomy, and bariatric surgery, and because it is a simple and safe block, it is gaining increasing acceptance in daily practice for the treatment of chronic and acute pain. The aim of postoperative analgesia management is to provide effective analgesia by using multimodal techniques, thus reducing opioid consumption and related complications, providing early mobilization and shorter hospital stay, and increasing patient comfort.

DETAILED DESCRIPTION:
Once the effectiveness of the Erector Spinae Plane Block has been demonstrated in patients undergoing robotic colorectal surgery, it will be implemented routinely in our clinic, aiming to reduce postoperative narcotic analgesic consumption, protect patients from narcotic analgesic side effects, facilitate early patient mobilization, shorten hospital stays, and increase patient comfort.

Because no additional procedures or medications were administered to patients outside of routine procedures, no additional risks are anticipated.

Pain is a subjective symptom, and to minimize interpatient variability, it will be assessed using the Numeric Rating Scale (NRS), a standardized scale.

The Postoperative Nausea Vomiting Impact Scale Score will be used to assess postoperative nausea and vomiting.

All volunteers participating in the study, whether or not a block is applied, will receive intravenous analgesia postoperatively using patient-controlled analgesia devices containing 4 mg/ml tramadol, with no basal infusion, a lockout time of 30 minutes, a bolus dose of 3 ml, and no baseline infusion. Data on the time of patients' first analgesic needs, the total number of analgesic requests and at what time, and the total tramadol dose administered will be obtained and recorded from the PCA devices.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Male and female gender
* Ages 18-75
* Malignant patients undergoing robotic colorectal surgery

Exclusion Criteria:

* ASA>III
* Coagulopathy
* Morbid obesity
* History of chronic analgesic use
* Data loss due to limited cooperation during NRS follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Total tramadol consumption in the first 24 hours after surgery | 24 hours
  Effect of ESPB on total tramadol consumption in the first 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative Resting Numerical Rating Scale (NRS) scores | 72 hours
  Postoperative resting Numerical Rating Scale (NRS) scores in 72 hours (minimum 0 - maximum 10)
Postoperative Deep Breathing/Coughing Numerical Rating Scale (NRS) scores | 72 hours
  Postoperative deep breathing/coughing Numerical Rating Scale (NRS) scores in 72 hours (minimum 0 - maximum 10)
Postoperative nausea and vomiting | 24 hours
  Evaluation of the frequency and severity of postoperative nausea and vomiting between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Burcu İzgi Duman, MD, Principal Investigator — Basaksehir Cam ve Sakura State Hospital
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identifying, formatting and transferring data into a standardized, usable electronic format can be time-consuming.